CLINICAL TRIAL: NCT05826236
Title: Effects of Joint Pressure Stimuli on Quadriceps Strength and Neuromuscular Activity in Patients With Knee Ostearthritis
Brief Title: Knee Pressure Stimuli on Quadriceps Strength in Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: CLF22/05
Record Dates: First submitted 2023-04-07; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis; Muscle Weakness
MeSH Terms: conditions — Osteoarthritis, Knee; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with knee osteoarthritis: Periarticular knee compression using a sphygmomanometer.
  Interventions: Device: Periarticular compression
- Healthy subjects: Periarticular knee compression using a sphygmomanometer.
  Interventions: Device: Periarticular compression

INTERVENTIONS:
Device: Periarticular compression — Periarticular knee compression using a sphygmomanometer.

SUMMARY:
The study aims at investigating the effects of a periarticular knee pressure stimulation on quadriceps strength and neuromuscular activity in subjects with knee ostearthritis.

Twenty-five patients with end-stage knee osteoarthritis and and twenty-five age-matched healthy subjects will be enrolled. All participants will be asked to performed isometric maximal voluntary knee extension tasks with three different pressure stimuli in terms of intensity (0 mmHg, 60 mmHg, 120 mmHg) around the knee using a sphygmomanometer. Peak force and root-mean-square peak of rectus femoris, vastus medialis, and vastus lateralis will be collected.

DETAILED DESCRIPTION:
The study aimed at assessing the effects of a periarticular pressure stimulation of the knee joint on quadriceps strength and neuromuscular activity in patients with end-stage knee osteoarthritis.

Twenty-five patients with end-stage knee osteoarthritis and and twenty-five age-matched healthy subjects will be enrolled. Participants will seat on a dynamometer chair (BAR, OTBioelettronica, Italy) with hips and knees at 90 degrees and 30 degrees of flexion, respectively. Participants will perform six maximal voluntary knee extension tasks with three different pressure stimuli in terms of intensity (0 mmHg, 60 mmHg, 120 mmHg) around the knee using a sphygmomanometer. Two maximum voluntary contractions interspaced by 3 minutes of rest will be performed for each pressure level, and the peak force (N) will be collected and normalized for the highest value during the three conditions. Moreover, root-mean-square peak (RMS-peak) of rectus femoris, vastus medialis, and vastus lateralis will be recorded using bipolar surface electromyography electrodes (FREEEMG, BTS, Italy). The RMS-peak of each muscle will be normalized for its highest value among the three conditions (nRMS-peak) and used as index of neuromuscular activity.

ELIGIBILITY:
Inclusion Criteria:

* End-stage knee osteoarthritis
* Age between 40 and 80 years
* at least 0-90° of knee range of motion along the sagittal plane

Exclusion Criteria:

* Cognitive impairments or psychiatric disorders
* Concomitant neurological, orthopedic, cardiovascular disorders
* Lower limb orthopedic surgery or traumatic events in the previous year

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with end-stage knee osteoarthritis with the aforementioned eligibility criteria and age-matched healthy subjects with the same criteria except "end-stage knee osteoarthritis".
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Peak Force | Baseline (0mmHg), 3 minute after baseline (60mmHg) and 6 minutes after baseline (120mmHg)
  Changes in strength during a maximal voluntary contraction using 0mmHg, 60mmHg or 120mmHg of compression intensity.

SECONDARY OUTCOMES:
Changes in Root Mean Square peak | Baseline (0mmHg), 3 minute after baseline (60mmHg) and 6 minutes after baseline (120mmHg)
  Changes in neuromuscular activity during a maximal voluntary contraction using 0mmHg, 60mmHg or 120mmHg of compression intensity.

IPD SHARING:
Plan to Share IPD: No